CLINICAL TRIAL: NCT01249430
Title: A Phase 1 Study of Azacitidine in Combination With MEC (Mitoxantrone, Etoposide, Cytarabine) in Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: Azacitidine in Combination With Mitoxantrone, Etoposide Phosphate, and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02554; NCI-2011-02554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000689575; OSU-10093; OSU 10093; 8803 (Other: Ohio State University Comprehensive Cancer Center); 8803 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Cytarabine; etoposide phosphate; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (azacitidine, mitoxantrone, etoposide, cytarabine) (Experimental): Patients receive azacitidine IV over 30 minutes on days 1-8 and mitoxantrone hydrochloride IV over 10 minutes, etoposide phosphate IV over 30-60 minutes, and cytarabine IV over 6 hours on days 3-8. Treatment continues for 1 course in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Cytarabine; Drug: Etoposide Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of azacitidine when given together with mitoxantrone, etoposide phosphate, and cytarabine in treating patients with acute myeloid leukemia that has returned after a period of improvement or does not respond to treatment. Azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as mitoxantrone, etoposide phosphate, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Azacitidine may help mitoxantrone, etoposide phosphate, and cytarabine work better by making cancer cells more sensitive to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose of azacitidine (5-azaC) when combined with mitoxantrone hydrochloride (mitoxantrone), etoposide phosphate (etoposide), and cytarabine (MEC) as salvage chemotherapy in patients with relapsed or refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To define the qualitative and quantitative toxicities of 5-azaC with MEC in combination with regard to organ specificity, time course, predictability, and reversibility.

II. To document the rate of complete remission (CR) and CR with incomplete blood count recovery (CRi) for this combination of agents as well as overall survival, relapse-free survival, and event-free survival.

III. To evaluate the pharmacokinetics of 5-azaC when given in combination with MEC in patients enrolled on this study.

IV. To measure R2 downregulation, including changes in R2 target, AraCTP, and dNTP/NTP pools, of 5-azaC in combination with MEC and correlate these pharmacodynamic endpoints with clinical response.

VI. To evaluate hypomethylation, including DMNT1 expression, Sp1 expression, global deoxyribonucleic acid (DNA) methylation, gene expression profiling, and micro ribonucleic acid (RNA) expression profiling, of 5-azaC when given in combination with MEC and correlate these pharmacodynamic changes with clinical response.

OUTLINE: This is a dose-escalation study of azacitidine.

Patients receive azacitidine intravenously (IV) over 30 minutes on days 1-8 and mitoxantrone hydrochloride IV over 10 minutes, etoposide phosphate IV over 30-60 minutes, and cytarabine IV over 6 hours on days 3-8. Treatment continues for 1 course in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed or refractory acute myeloid leukemia (AML) according to 2008 World Health Organization (WHO) classification; must have failed at least one cycle of induction chemotherapy or relapsed after achieving a complete remission following induction chemotherapy; patients with prior autologous or allogeneic stem cell transplant are permitted
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months for any comorbid conditions
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 mg/dL
* Left ventricular ejection fraction >= 40%
* Ability to understand and the willingness to sign a written informed consent document
* Patients must have recovered from the non-hematologic toxicity of prior therapy to less than grade 2

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients receiving any other investigational agents or patients that have received any other investigational agents within 14 days of enrollment
* Patients with active central nervous system disease or with granulocytic sarcoma as sole site of disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacitidine, mannitol, or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients with active infection are permitted to enroll provided that the infection is under control; myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any echocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with azacitidine
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01-20 (Actual); Primary Completion 2013-05-24 (Actual); Study Completion 2013-05-24 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of azacitidine when combined with salvage chemotherapy (mitoxantrone hydrochloride, etoposide, and cytarabine [MEC]) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to day 42
  Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Clinical response according to the International Working Group criteria | Up to day 42
  Responses will be summarized by simple descriptive summary statistics delineating complete and lesser responses as well as stable and progressive disease.
Qualitative and quantitative toxicities of azacitidine in combination with (mitoxantrone hydrochloride, etoposide, and cytarabine [MEC]) | Up to 30 days post-therapy
  Graded according to NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Walker, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States